CLINICAL TRIAL: NCT04064749
Title: Developing and Testing a Brief Intervention for Problem Gambling in Credit Counseling
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: National Center for Responsible Gaming (Other)
Responsible Party: Principal Investigator, Jodi Jacobson Frey, Associate Professor, University of Maryland, Baltimore
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: HP-00084892
Record Dates: First submitted 2019-08-12; First posted 2019-08-22 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2024-04

CONDITIONS: Gambling Problem
MeSH Terms: interventions — Crisis Intervention

STUDY DESIGN:
Intervention Model Description: The Screening, Brief Intervention and Referral to Treatment (SBIRT) model provides the underlying structure for the proposed brief intervention. SBIRT interventions utilize a combination of brief educational approaches (i.e., information about risks of use) combined with motivational interviewing techniques designed to enhance motivation to make a change in a target behavior.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Participants will receive screening (i.e. services as usual) provided by a national credit counseling program.
- Intervention (Experimental): Participants will receive screening services provided by the credit counseling program plus added brief intervention services by University of Maryland School of Social Work (UMSSW). Added intervention services include: 1) feedback about the individual's gambling, and 2) text messages to support the individual.
  Interventions: Behavioral: Text messages

INTERVENTIONS:
Behavioral: Text messages — The brief intervention includes providing feedback on the individual's gambling score; providing an educational fact about the relationship between problem gambling and financial well-being; talking with the individual about the 'pros' and 'cons' of gambling with suggested strategies that could potentially reduce their gambling behaviors; and concluding with an action oriented closing question. Participants in the intervention group will also receive up to five text messages a week for one month.
  Other Names: Brief intervention
  Arms: Intervention

SUMMARY:
This study will implement a brief intervention with text messaging and will test its effectiveness in reducing gambling behavior and improving financial well-being among credit counseling clients who seek services.

Financial counseling organizations provide a community-based environment for screening and brief intervention for gambling-related problems as gambling problems are fundamentally about financial losses. The study holds the promise of expanding brief interventions for gambling to individuals outside the health care system and in so doing, help those at-risk who do not present for formal treatment.

DETAILED DESCRIPTION:
The randomized control trial is designed to test the effectiveness of a unique brief intervention for at-risk gambling within a national financial counseling organization. Individuals who call the program for credit counseling and financial support will be asked a brief screen for problem gambling by a trained financial advocate (i.e. credit counselor). Individuals who are eligible for the study will be provided with information about the study by their financial advocate and asked if they would be willing to have a researcher at University of Maryland School of Social Work (UMSSW) contact them to tell them more about information about the study and review informed consent.

If the person wants to learn more about the study, a member of the research team at UMSSW will contact the individual, who will review the informed consent with the individual and answer questions. After obtaining their consent, the researcher will randomize the individual to either Group 1 (control) or Group 2 (intervention). A randomization matrix will be prepopulated in advance so that the researcher will assign the individual based on the next group assignment. If the individual is randomly assigned to Group 1, the researcher will proceed by asking the baseline/Time 1 interview questions. They will not receive any additional intervention.

If the individual is randomly assigned to Group 2, the researcher will proceed by providing the brief intervention. The brief intervention includes providing feedback on the individual's gambling score; providing an educational fact about the relationship between problem gambling and financial well-being; talking with the individual about the 'pros' and 'cons' of gambling with suggested strategies that could potentially reduce their gambling behaviors; and concluding with an action oriented closing question. Following the intervention, the researcher will then administer the baseline/Time 1 structured interview questions.

For individuals who are assigned to the intervention group, they will also receive text messages. The researchers will send text messages via pre-programmed, automated mode to the client. Participants will receive up to five messages a week, and messages will be delivered at times when gambling may be higher, such as weekend afternoons and evenings. Text messages will be sent following baseline for one month, through the end of T2 (30-day post screening).

Individuals who agree to participate in the study and who are randomized to either group (control or intervention) will complete three phone interviews by phone that inquire about gambling behaviors, financial well-being, and mental health-seeking behavior. Phone interviews will be administered at baseline (Time 1), 30 days (Time 2), and 90 days (Time 3) following consent. The credit counseling program will also provide data from their initial evaluation and screening from their records on individuals who take part in the intervention (e.g., sociodemographic variables, financial information about assets and debt, and the results of the gambling screen).

ELIGIBILITY:
Inclusion Criteria:

* over age 18;
* can speak and understand English;
* called credit counseling program for services; and
* scored at risk for problem gambling on the questions asked by the financial advocate

Exclusion Criteria:

* younger than 18
* cannot speak and understand English
* did not call credit counseling program for services; and
* did not score at risk for problem gambling on the questions asked by the financial advocate

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2021-08-28 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Brief Problem Gambling Screen | screener asked at baseline when individuals call in to Consumer Credit Counseling Services of Maryland
  The Brief Problem Gambling Screen is a 5-item screening measure ideal for assessing at-risk, problem, or pathological gamblers in both clinical settings and population research. Through yes/no questions, this scale employs three behavior items, one motivation item, and one consequences item with positive endorsement of one or more items indicating a problem with gambling.
The South Oaks Gambling Screen (SOGS) | baseline
  The South Oaks Gambling Screen (SOGS) will be administered at baseline to estimate the level of lifetime gambling risk among participants in the study. Scores on the SOGS are determined by scoring one point for each question that shows the "at risk" response indicated and adding the total points. A score of 0 means No problem with gambling; scores of 1-4 indicate Some problems with gambling; and scores of 5 or more indicate Probable pathological gambler.
Gambling Symptoms Assessment Scale (GSAS) - change is being assessed over time | baseline, Time 2 (30 days post randomization), Time 3 (90 days post randomization)
  Gambling Symptoms Assessment Scale (GSAS) measures self-rated gambling severity using 12 Likert scale items. The GSAS asks the respondent about a variety of gambling-related problems over a fairly brief recall period (one-week). The scale's response options range from none to extreme or constant. In scoring the GSAS each item is scored on a 5-point scale from 0 (no symptoms) to 4 (extreme symptoms). The total score ranges from 0 to 48 with higher scores indicating greater gambling problems.
The Financial Well-Being Assessment Scale - change is being assessed over time | baseline, Time 2 (30 days post randomization), Time 3 (90 days post randomization)
  The Financial Well-Being Assessment Scale was developed by the Consumer Financial Protection Bureau and is a reliable and valid measure of perceived financial well-being. The measure contains ten Likert scale items with response options ranging from completely or always to not at all or never. This instrument will provide a precise estimate of financial well-being at each time point with lower scores indicating lower financial well-being.
Mental Help Seeking Intention Scale - change is being assessed over time | baseline, Time 2 (30 days post randomization), Time 3 (90 days post randomization)
  The Mental Help Seeking Intention Scale is a three-item measure which assesses an individual's intent to seek help for a mental health problem. Response options range from extremely likely or strongly agree to extremely unlikely or strongly disagree.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Maryland Baltimore, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No